CLINICAL TRIAL: NCT02740153
Title: Comparative Effectiveness of Therapy in Rare Diseases: Liver Transplantation vs. Conservative Management of Urea Cycle Disorders
Brief Title: PCORI Urea Cycle Disorder Study
Status: Completed | Type: Observational
Sponsor: Children's National Research Institute (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Patient-Centered Outcomes Research Institute (Other); George Washington University (Other); The National Urea Cycle Disorders Foundation (Unknown); Studies of Pediatric Liver Transplantation (Unknown)
Responsible Party: Principal Investigator, Nicholas Ah Mew, MD, Children's National Research Institute
Other Study IDs: 7282
Record Dates: First submitted 2016-03-29; First posted 2016-04-15 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Urea Cycle Disorders
MeSH Terms: conditions — Urea Cycle Disorders, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Urea Cycle Disorder with Liver Transplant: * Age 18 and under
  * Diagnosed with the following Neonatal-type urea cycle disorders: CPSD, OTCD, ASD or ALD
  * History of liver transplant
  Interventions: Other: No Intervention Given
- Urea Cycle Disorder without Transplant: * Age 18 and under
  * Diagnosed with the following Neonatal-type urea cycle disorders: CPSD, OTCD, ASD or ALD
  * No history of liver transplant, managed medically
  Interventions: Other: No Intervention Given

INTERVENTIONS:
Other: No Intervention Given

SUMMARY:
Urea cycle disorders (UCD) are genetic disorders caused by the liver's inability to break down ammonia from proteins; ammonia then accumulates and is toxic to the brain. UCD cause brain damage and intellectual and developmental disabilities and even death.

Treatment for UCD is either conservative management which involves a low-in-protein diet, drugs, and amino acid supplements or liver transplantation; each carries their own risks.

This study aims to help patients to make the decision about different management alternatives by providing them with scientific information that is currently lacking.

Aim 1 of this study will compare survival, neurocognitive function, and patient-reported quality of life.

DETAILED DESCRIPTION:
Urea cycle disorders (UCD) are genetic disorders caused by the liver's inability to break down ammonia from proteins; ammonia then accumulates and is toxic to the brain. UCD cause brain damage and intellectual and developmental disabilities and even death.

Treatment involves a special diet low in protein, drugs that help metabolize ammonia and amino acid supplements (conservative management). Many patients and families choose liver transplantation rather than conservative treatment; both alternatives are effective in reducing or normalizing blood ammonia. While liver transplantation eliminates the ammonia problem, conservative management does so only temporarily and in many patients, blood ammonia can rise during an infection.

The long-term objective of this study is to help patients make decisions about management alternatives (conservative vs. liver transplantation) by providing them with scientific information that is currently lacking. The questions the investigators will address are:

1. What is the disease's risk of mortality and illness in the two treatment approaches?
2. What can parents expect in terms of the development of their child and his/her school performance?
3. What are the expected effects of each treatment on short-term and long-term quality of life?

The investigators will use statistical methods to compare numbers or percentages of survival, illness, psychological testing for IQ, executive function, memory, behaviors, and quality of life among patients that choose conservative management and those who have chosen liver transplantation. Some of this information is already being collected by the Urea Cycle Disorders Consortium (UCDC) in 14 metabolic clinics (11 of them in the US) as part of its long-term follow-up study. To ensure that the information the investigators analyze is representative of the UCD patient population in the US, the investigators will also obtain data from the Studies of Pediatric Liver Transplantation (SPLIT) registry, which collects information about children who undergo liver transplantation for many different diseases (including UCD).

The National Urea Cycle Disorders Foundation (NUCDF) and the Patients' Research Working Group collaborated with the clinical investigators to design this research and to ensure that it that it covers the questions that are most important to patients and their families. The results of this study will be disseminated to patients, their doctors, and clinical staff so they receive current, validated information before making a decision about the best treatment for them.

ELIGIBILITY:
Inclusion Criteria:

Aim 1 (UCD patients):

* Age 18 and under
* Diagnosed with the following Neonatal-type urea cycle disorders:
* CPSD, OTCD, ASD or ALD, as defined as follows:

  * Diagnosis of CPS I deficiency, defined as decreased (less than 20 % of control) CPS I enzyme activity in liver, and/or an identified pathogenic mutation, and/or hyperammonemia and first-degree relative meets at least one of the criteria for CPS I deficiency
  * Diagnosis of OTC deficiency, defined as the identification of a pathogenic mutation, and/or less than 20% of control of OTC activity in the liver, and/or elevated urinary orotate (greater than 20 uM/mM) in a random urine sample or after allopurinol challenge test, and/or hyperammonemia and first degree relative meets at least one of the criteria for OTC deficiency
  * Diagnosis of AS deficiency (Citrullinemia), defined as a greater than or equal to 10-fold elevation of citrulline in plasma, and/or decreased (less than 20% of control) AS enzyme activity in cultured skin fibroblasts or other appropriate tissue, and/or identification of a pathogenic mutation in the AS gene, and/or hyperammonemia and first degree relative meets at least one of the criteria for AS Deficiency
  * Diagnosis of AL deficiency (Argininosuccinic Aciduria, ASA), defined as the presence of argininosuccinic acid in the blood or urine, and/or decreased (less than 20% of control) AL enzyme activity in cultured skin fibroblasts or other appropriate tissue, and/or identification of a pathogenic mutation in the AL gene, and/or hyperammonemia and first degree relative meets at least one of the criteria for AL Deficiency
* Willing to participate in at least 1 neurocognitive assessment and 1 quality of life assessment
* Permit access to medical records and medical providers

Exclusion Criteria:

Aim 1:

* Rare and unrelated comorbidities (e.g., Down's syndrome, intraventricular hemorrhage in the newborn period, and extreme prematurity)

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population for Aim 1 includes children aged 18 and younger who are diagnosed with one of the following Neonatal-type urea cycle disorders: CPSD, OTCD, ASD, or ALD. Participants will come from children's hospitals and pediatric clinics that treat urea cycle disorders throughout the country.
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mendel Tuchman, MD, Study Chair — Children's National Research Institute; Nicholas Ah Mew, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Childrens Research Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Urea Cycle Disorder Consortium registry study and were recruited from UCDC member hospitals. Recruitment began in April 2016 and ended in April 2019.
Pre-assignment Details: No pre-assignment details, this was not an intervention study.
Groups:
- Urea Cycle Disorder With Liver Transplant: * Age 18 and under
  * Diagnosed with the following Neonatal-type urea cycle disorders: CPSD, OTCD, ASD or ALD, as defined as follows:
  History of liver transplant.
  No intervention given.
- Urea Cycle Disorder Without Transplant: * Age 18 and under
  * Diagnosed with the following Neonatal-type urea cycle disorders: CPSD, OTCD, ASD or ALD, as defined as follows:
  No history of liver transplant, managed conservatively with medication and diet.
  No intervention given.
Period: Overall Study
Arm/Group | Urea Cycle Disorder With Liver Transplant | Urea Cycle Disorder Without Transplant
Started | 101 | 86
Completed | 101 | 86
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Urea Cycle Disorder With Liver Transplant: * Age 18 and under
  * Diagnosed with the following Neonatal-type urea cycle disorders: CPSD, OTCD, ASD or ALD, as defined as follows:
  No Intervention Given
  History of liver transplant
- Urea Cycle Disorder Without Transplant: * Age 18 and under
  * Diagnosed with the following Neonatal-type urea cycle disorders: CPSD, OTCD, ASD or ALD, as defined as follows:
  No Intervention Given
  No history of liver transplant
- Total: Total of all reporting groups
Arm/Group | Urea Cycle Disorder With Liver Transplant | Urea Cycle Disorder Without Transplant | Total
Number analyzed (Participants) | 101 | 86 | 187
Age, Customized [Count of Participants; unit: Participants] — Population: Number analyzed in rows is the same as overall for comparison of Aim 1 arms (liver transplant versus medical management)
  Participants
    <6 Months | 20 | 28 | 48
    6-12 Months | 29 | 10 | 39
    1-5 Years | 38 | 35 | 73
    5-10 Years | 10 | 10 | 20
    >10 Years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 67 | 53 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 11 | 28
  Not Hispanic or Latino | 77 | 62 | 139
  Unknown or Not Reported | 7 | 13 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: This aspect of Aim 1 is prospective by design based on selection by exposure (liver transplant or medical managed) evaluating the clinical outcomes of subjects with urea cycle disorders.
Time Frame: 436 person years in the Liver Transplant Group and 386 person-years in the Without Transplant Group
Population: Treatment-related effects on mortality
Measure: Number (95% Confidence Interval); unit: participant per 1000 person-years
Groups:
- Urea Cycle Disorder Without Transplant: * Age 18 and under
  * Diagnosed with the following Neonatal-type urea cycle disorders: CPSD, OTCD, ASD or ALD, as defined as follows:
  No Intervention Given
  No history of liver transplant, UCD managed conservatively through medical management
Arm/Group | Urea Cycle Disorder With Liver Transplant | Urea Cycle Disorder Without Transplant
Number analyzed (Participants) | 101 | 86
participant per 1000 person-years | 18.4 [9.2 to 36.7] | 20.7 [10.4 to 41.4]

2. Primary Outcome: Neurocognitive Function: Full-Scale IQ
Description: Neuropsychological tests were based on age-matched norms for the specific test used. All neurocognitive scores have been standardized to the following: norm, mean of 100, and sd of 15. In all tests higher scores are interpreted as higher functions. The WPPSI and WASI were combined to create a single measure of Full-Scale IQ.
  Full-Scale IQ
  * Wechsler Preschool and Primary Scales of Intelligence, 4th edition (WPPSI-IV: Children 3-5 years of age)
  * Wechsler Abbreviated Scales of Intelligence, 1st and 2nd editions (WASI-I & II: Persons 6+ years of age)
Time Frame: Neuropsychological testing was conducted once for each patient at baseline during the study on age-matched norms for the specific test used.
Population: * Full Scale IQ
  * WPPSI - Children 3-5 years of age
  * WASI - Persons 6+ years of age
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Urea Cycle Disorder Without Transplant: * Age 18 and under
  * Diagnosed with the following Neonatal-type urea cycle disorders: CPSD, OTCD, ASD or ALD, as defined as follows:
  No Intervention Given
  No history of liver transplant. UCD managed conservatively with medical intervention.
Arm/Group | Urea Cycle Disorder With Liver Transplant | Urea Cycle Disorder Without Transplant
Number analyzed (Participants) | 15 | 25
score on a scale | 80.1 [67.5 to 92.7] | 82 [73.5 to 90.6]

3. Primary Outcome: Total Quality of Life
Description: Quality of life assessments are self-reported by participating patients or by their parent/caretaker using the following reports:
  Pediatric Family Impact (PedsQL), Version 4 is reported as a total score
  All were scored on a 0-100 scale. Higher scores indicated a better health-related quality of life
Time Frame: Quality of life testing was conducted and reported at baseline for each patient during the study.
Population: Patient/family reported quality of life using PedsQL quality of life measuremet tool (version 4)
Measure: Mean (95% Confidence Interval); unit: score on a scale of 0-100
Groups:
- Urea Cycle Disorder Without Transplant: * Age 18 and under
  * Diagnosed with the following Neonatal-type urea cycle disorders: CPSD, OTCD, ASD or ALD, as defined as follows:
  No Intervention Given
  No history of liver transplant. UCD managed conservatively through medical intervention.
Arm/Group | Urea Cycle Disorder With Liver Transplant | Urea Cycle Disorder Without Transplant
Number analyzed (Participants) | 23 | 16
score on a scale of 0-100 | 69.8 [60.9 to 78.7] | 55.6 [44.7 to 66.5]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected on enrolled patients every month throughout the study until study completion.
Description: Adverse event definitions do not differ from the clinicaltrials.gov definitions.
Arm/Group | Urea Cycle Disorder With Liver Transplant | Urea Cycle Disorder Without Transplant
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/86
Other Adverse Events (participants affected / at risk) | 0/101 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT02740153/Prot_SAP_000.pdf